CLINICAL TRIAL: NCT07214922
Title: A Phase I, Open-Label Study of the Relative Bioavailability of Evobrutinib Tablet Manufacturing Batches in Healthy Participants
Brief Title: Relative Bioavailability of Evobrutinib Tablet Batches
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200527_0131; 2022-002755-19 (EudraCT Number)
Record Dates: First submitted 2025-10-08; First posted 2025-10-09 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Evobrutinib; Pharmacokinetics; Relative Bioavailability; Crossover
MeSH Terms: interventions — evobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Evobrutinib: Treatment Sequence 1: ABCD (Experimental): Participants will receive single oral dose of Treatment A on Day 1 in period 1, followed by single oral dose of Treatment B on Day 3 in period 2, followed by Treatment C on Day 5 in period 3 and followed by single oral dose of Treatment D on Day 7 under fasted condition in period 4. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Evobrutinib: Treatment Sequence 2: BDAC (Experimental): Participants will receive single oral dose of Treatment B on Day 1 in period 1, followed by single oral dose of Treatment D on Day 3 in period 2, followed by Treatment A on Day 5 in period 3 and followed by single oral dose of Treatment C on Day 7 under fasted condition in period 4. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Evobrutinib: Treatment Sequence 3: CADB (Experimental): Participants will receive single oral dose of Treatment C on Day 1 in period 1, followed by single oral dose of Treatment A on Day 3 in period 2, followed by Treatment D on Day 5 in period 3 and followed by single oral dose of Treatment B on Day 7 under fasted condition in period 4. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D
- Evobrutinib: Treatment Sequence 4: DCBA (Experimental): Participants will receive single oral dose of Treatment D on Day 1 in period 1, followed by single oral dose of Treatment C on Day 3 in period 2, followed by Treatment B on Day 5 in period 3 and followed by single oral dose of Treatment A on Day 7 under fasted condition in period 4. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D

INTERVENTIONS:
Drug: Treatment A — Participants will receive single dose of Treatment A in treatment period 1, 2, 3 or 4 under fasted conditions.
  Other Names: Evobrutinib
Drug: Treatment B — Participants will receive single dose of Treatment B in treatment period 1, 2, 3 or 4 under fasted conditions.
  Other Names: Evobrutinib
Drug: Treatment C — Participants will receive single dose of Treatment C in treatment period 1, 2, 3 or 4 under fasted conditions.
  Other Names: Evobrutinib
Drug: Treatment D — Participants will receive single dose of Treatment D in treatment period 1, 2, 3 or 4 under fasted conditions.
  Other Names: Evobrutinib

SUMMARY:
The main purpose of the study is to compare the Pharmacokinetics (PK), safety and tolerability of different manufacturing batches of M2951 tablet formulation relative to a reference batch under fasted conditions in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection, or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Participants who have a body weight within 50.0 and 100.0 kilogram (kg) (inclusive) and Body Mass Index within the range 19.0 and 30.0 kg/ meter square (m2) (inclusive)
* Female participant who agrees to use appropriate contraception and barrier methods.
* Male participants: No contraception needed
* Participants who are capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and this protocol
* Participants who are stable non-smokers for at least 3 months preceding Screening
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with history or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, musculoskeletal, genitourinary, immunological, dermatological, connective tissue, psychiatric (due to rare risk of hallucinations, agitation and activation of psychosis), and other diseases or disorders, and epilepsy, as determined by medical evaluation
* Participants with diagnosis of hemochromatosis, Wilson´s disease, alpha 1 antitrypsin deficiency, or any other chronic liver disease including Gilbert's disease will be excluded from the study
* Participants with prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to the first administration of study intervention
* Participants with history of any malignancy
* Participants with history of seizures
* Participants with history of pharmacologically treated psychiatric disease
* Participants with history of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to the first administration of study intervention
* Participants with history of shingles within 12 months prior to Screening
* Participants with history of drug hypersensitivity
* Participants with history of residential exposure to tuberculosis, or a positive QuantiFERON® test within 4 weeks prior to or at the time of Screening
* Participants positive for

  1. hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or Human Immunodeficiency Virus (HIV) I and II tests at Screening
  2. severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening and Day -1
* Participants with any condition, including findings in the laboratory tests, medical history (example heart failure, hypokalemia, family history of Long QT Syndrome), or other Screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation
* Participants with history of administration of live vaccines or live-attenuated virus vaccines within 3 months prior to Day 1.
* Participants with history of administration of other types of vaccines is allowed until 14 days before the first administration of study intervention, thereafter it is prohibited until the end of the study.
* Participants with Moderate or strong inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4)/5 or Pgp within 4 weeks prior to the first administration of study intervention
* Participants with use of any prescribed medicine or over-the-counter drug or dietary supplement, including herbal remedies, vitamins, and minerals, antacids and dietary supplements such as fish oils within 2 weeks or 5 times the half-life of the respective drug, whichever is longer, prior to the first administration of study intervention
* Participants with use of any investigational drug in any clinical study within 60 days prior to Day 1 administration, or have used an experimental monoclonal antibody within the past 1 year prior to Day 1, or have participated in a study evaluating a Bruton Tyrosine Kinase (BTK) inhibitor within 60 days, or are on extended follow-up in a clinical study, even if last administration of a study intervention was more than 60 days ago, or 5 half-lives of the investigational drug, whichever is longer, prior to the first administration of study intervention
* Participants with a medical history and physical examination results that include any ongoing clinically relevant findings as judged by the Investigator
* Participants with clinically relevant findings (excluding minor, not clinically relevant excursions from normal ranges, as judged by the Investigator) at Screening in biochemistry, hematology, coagulation, and urinalysis examinations for the age of the participant, as judged by the Investigator:

  * Alanine aminotransferase, aspartate aminotransferase: above upper limit of normal (ULN)
  * Creatinine: above normal limits
  * Absolute lymphocyte count, absolute neutrophil count: below limit of reference range.
  * Amylase and lipase above normal ranges; minor deviations are allowed, if not clinically relevant.
* Participants with estimated glomerular rate (eGFR) according to the Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation (2009) < 90 milliliters/minute(mL/min) at Screening. In case of a borderline result between ≥ 80 and < 90 mL/min, Cystatin C will be determined in addition, and the participant will only be included if the Cystatin C value is below the upper limit of normal
* Participants with semi-supine systolic blood pressure > 140 mmHg or < 90 millimeters of mercury (mmHg), diastolic blood pressure > 90 mmHg or < 50 mmHg, and pulse rate > 90 or < 50 beats per minute (bpm) at Screening.
* Participants with consumption of alcohol from 48 hours prior to first administration of study intervention.
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/
- See also: Medical Information Location Map - Med Info Contacts — http://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Treatment A-B-C-D: Participants received single oral dose of reference treatment (treatment A) of Evobrutinib (45 milligrams [mg]) on Day 1 in period 1, followed by single oral dose of lower dissolution bound batch (treatment B) of Evobrutinib (45 mg) on Day 3 in period 2, followed by single oral dose of upper dissolution bound batch (treatment C) of Evobrutinib (45 mg) on Day 5 in period 3 and followed by single oral dose of hammer milled batch (treatment D) of Evobrutinib (45 mg) on Day 7 under fasted condition in period 4. A washout period of 48 hours was maintained between 4 treatment periods.
- Sequence 2: Treatment B-D-A-C: Participants received single oral dose of lower dissolution bound batch (treatment B) of Evobrutinib (45 mg) on Day 1 in period 1, followed by single oral dose of hammer milled batch (treatment D) of Evobrutinib (45 mg) on Day 3 in period 2, followed by single oral dose of reference treatment (treatment A) of Evobrutinib (45 (mg) on Day 5 in period 3 and followed by single oral dose of upper dissolution bound batch (treatment C) of Evobrutinib (45 mg) on Day 7 under fasted condition in period 4. A washout period of 48 hours was maintained between 4 treatment periods.
- Sequence 3: Treatment C-A-D-B: Participants received single oral dose of upper dissolution bound batch (treatment C) of Evobrutinib (45 mg) on Day 1 in period 1, followed by single oral dose of reference treatment (treatment A) of Evobrutinib (45 (mg) on Day 3 in period 2, followed by single oral dose of hammer milled batch (treatment D) of Evobrutinib (45 mg) on Day 5 in period 3 and followed by single oral dose of lower dissolution bound batch (treatment B) of Evobrutinib (45 mg) on Day 7 under fasted condition in period 4. A washout period of 48 hours was maintained between 4 treatment periods.
- Sequence 4: Treatment D-C-B-A: Participants received single oral dose of hammer milled batch (treatment D) of Evobrutinib (45 mg) on Day 1 in period 1, followed by single oral dose of upper dissolution bound batch (treatment C) of Evobrutinib (45 mg) on Day 3 in period 2, followed by single oral dose of lower dissolution bound batch (treatment B) of Evobrutinib (45 mg) on Day 5 in period 3 and followed by single oral dose of reference treatment (treatment A) of Evobrutinib (45 (mg) on Day 7 under fasted condition in period 4. A washout period of 48 hours was maintained between 4 treatment periods.
Period: Overall Study
Arm/Group | Sequence 1: Treatment A-B-C-D | Sequence 2: Treatment B-D-A-C | Sequence 3: Treatment C-A-D-B | Sequence 4: Treatment D-C-B-A
Started | 7 | 7 | 7 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — DROPPED OUT ON DAY 5; PRIVATE REASONS | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Treatment A-B-C-D | Sequence 2: Treatment B-D-A-C | Sequence 3: Treatment C-A-D-B | Sequence 4: Treatment D-C-B-A | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30 (5.6) | 37 (10.1) | 37 (12.8) | 35 (10.4) | 35 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 5 | 17
  Male | 3 | 2 | 4 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 6 | 7 | 7 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 7 | 7 | 7 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Evobrutinib
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: Pharmacokinetic (PK) Analysis Set was a subset of the Safety Analysis Set and included all participants who receive at least one dose of active investigational medicinal product (IMP) and provide at least one measurable post-dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour×nanogram per milliliter (h×ng/mL)
Groups:
- Treatment A: Participants received single dose of reference treatment (treatment A) of Evobrutinib (45 mg]) in treatment period 1, 2, 3 or 4 under fasted conditions.
- Treatment B: Participants received single dose of lower dissolution bound formulation (treatment B) of Evobrutinib (45 mg) in treatment period 1, 2, 3 or 4 under fasted conditions.
- Treatment C: Participants received single dose of upper dissolution bound formulation (treatment C) of Evobrutinib (45 mg) in treatment period 1, 2, 3 or 4 under fasted conditions.
- Treatment D: Participants received single dose of hammer milled formulation (treatment D) of Evobrutinib (45 mg) in treatment period 1, 2, 3 or 4 under fasted conditions.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
hour×nanogram per milliliter (h×ng/mL) | 198 (44.0) | 164 (45.1) | 207 (44.6) | 205 (38.3)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Evobrutinib
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
nanogram per milliliter (ng/mL) | 111 (69.9) | 84.5 (71.9) | 117 (62.6) | 121 (64.7)

3. Secondary Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events with onset date or worsening during the on-treatment period. TEAEs included both serious and non-serious TEAEs.
Time Frame: Up to 34 days
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
Participants | 2 | 1 | 2 | 5

4. Secondary Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs) by Severity
Description: The Investigator assessed the severity of each AE and SAE reported during the study and assign it to one of the following categories: Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities; Severe: An event that prevents normal everyday activities. Do not confuse an AE that is assessed as severe with a SAE. Severe is a category used to rate the intensity of an event; both AEs and SAEs can be assessed as severe.
Time Frame: Up to 34 days
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
Participants
  Mild | 2 | 0 | 0 | 4
  Moderate | 0 | 1 | 1 | 1
  Severe | 0 | 0 | 1 | 0

5. Secondary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure and Diastolic Blood Pressure
Description: Diastolic blood pressure and systolic blood pressure were measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline (Pre-dose), 2 hours post-dose
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
millimeters of mercury (mmHg)
  Systolic Blood Pressure | 0 (10.4) | -1 (7.3) | -1 (6.9) | -1 (7.0)
  Diastolic Blood Pressure | -1 (5.8) | -1 (5.8) | 0 (6.0) | -1 (4.7)

6. Secondary Outcome: Change From Baseline in Vital Signs: Temperature
Description: Temperature was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline (Pre-dose), 2 hours post-dose
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
degree Celsius | 0.2 (0.27) | 0.2 (0.34) | 0.0 (0.24) | 0.0 (0.27)

7. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate
Description: Pulse rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline (Pre-dose), 2 hours post-dose
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
beats per minute | -2 (8.5) | -1 (8.6) | -3 (8.3) | -2 (7.3)

8. Secondary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: Respiratory rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline (Pre-dose), 2 hours post-dose
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
breaths per minute | 0 (2.5) | -1 (2.0) | -1 (1.9) | -0 (2.0)

9. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) Parameter: Heart Rate
Description: Heart rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions
Time Frame: Baseline (Pre-dose), 2 hours post-dose
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
beats per minute | -4 (6.1) | -2 (4.0) | -2 (6.6) | -1 (4.7)

10. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) Parameter: RR Duration, QT Duration, QTcF Duration, PR Duration, QRS Duration
Description: RR Duration, QT Duration, QTcF Duration, PR Duration, QRS Duration was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline (Pre-dose), 2 hours post-dose
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
millisecond (msec)
  RR Duration | 52 (84.6) | 36 (61.3) | 44 (106.4) | 18 (70.3)
  QT Duration | 9 (10.9) | 6 (9.8) | 10 (10.7) | 4 (10.1)
  QTcF Duration | 1 (11.8) | 1 (9.5) | 4 (8.9) | 2 (8.7)
  PR Duration | -5 (7.8) | -1 (6.1) | -0 (8.0) | 0 (5.8)
  QRS Duration | -0 (4.9) | -1 (4.9) | 1 (4.8) | -1 (4.6)

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters
Description: Laboratory investigation included hematology, biochemistry and urinalysis. The number of participants with clinically significant changes from baseline in laboratory parameters were reported. Clinical significance was determined by the investigator.
Time Frame: Screening up to Day 8
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Evobrutinib
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification (LLOQ). Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h×ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
h×ng/mL | 194 (44.5) | 160 (46.3) | 204 (45.1) | 202 (39.2)

13. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Evobrutinib
Description: Time to reach the maximum observed plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
hours | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 2.00] | 1.00 [0.250 to 1.50] | 1.00 [0.500 to 2.00]

14. Secondary Outcome: Terminal Half Life (T1/2) of Evobrutinib
Description: Terminal half-life was calculated as log2 divided by lambda z. Lambda z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
hours | 1.64 [1.01 to 10.8] | 1.78 [1.05 to 13.7] | 1.72 [1.07 to 15.6] | 1.37 [0.982 to 5.41]

15. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Evobrutinib
Description: Apparent total body clearance of drug from plasma following extravascular administration, calculated as dose/AUC0-infinity for Evobrutinib.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
Liter per hour | 227 (44.0) | 275 (45.1) | 217 (44.6) | 219 (38.3)

16. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (VZ/f) of Evobrutinib
Description: Vz/f is defined as the apparent volume of distribution during the terminal phase following extravascular administration for Evobrutinib.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 27 | 27 | 27
Liters | 627 (84.1) | 843 (111.4) | 658 (89.2) | 522 (74.2)

17. Secondary Outcome: Relative Bioavailability Based on Area Under the Plasma Concentration Curve From Time Zero Extrapolated to Infinity [Frel(AUC0-inf)] of Evobrutinib (Treatment B, C and D) Compared to Evobrutinib Reference Treatment A
Description: Relative Bioavailability in percentage of each treatment (B, C, and D) in relation to the reference Treatment (A) was calculated as Frel = 100 multiplied by (AUC0-inf [treatment B, C, D]) multiplied by Dose [treatment A] divided by (AUC0-inf [treatment A]) multiplied by Dose [treatment B, C, D]. Treatment A to determine relative bioavailability.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose on Days 1, 3, 5 and 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percentage bioavailability
Arm/Group | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 26 | 26
percentage bioavailability | 84.0 [75.8 to 93.1] | 105 [98.1 to 112] | 106 [98.0 to 115]

ADVERSE EVENTS:
Time Frame: Up to 34 days
Groups:
- Treatment A: Participants received single dose of reference treatment (treatment A) of Evobrutinib (45 mg) in treatment period 1, 2,3 or 4 under fasted conditions.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 1/27 | 0/27
Other Adverse Events (participants affected / at risk) | 2/26 | 1/27 | 1/27 | 5/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=26) | Treatment B (N=27) | Treatment C (N=27) | Treatment D (N=27)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=26) | Treatment B (N=27) | Treatment C (N=27) | Treatment D (N=27)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT07214922/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT07214922/SAP_001.pdf